CLINICAL TRIAL: NCT02603250
Title: Evaluation of Hemoglobin Measurement Tools for Child Anemia Screening in Rwanda
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: University of Rwanda (Other)
Responsible Party: Sponsor
Other Study IDs: 703581-3
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-09

CONDITIONS: Anemia
Keywords: Anemia; Iron deficiency; noninvasive anemia screening
MeSH Terms: conditions — Anemia; Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Wicking: 50% of the 132 children enrolled in the study will have their Hb measured using the wicking method of HemoCue® 201+ blood collection.
- Gravity: 50% of the 132 children enrolled in the study will have their Hb measured using the gravity method of HemoCue® 201+ blood collection.

SUMMARY:
The purpose of this study is to evaluate the use of a noninvasive Hb device (Pronto® with DCI-mini™ sensors) as an accurate method for measuring Hb levels among children between 6 and 59 months against the standard reference hematology analyzer. The secondary purpose is to evaluate the accuracy of two HemoCue® Hb 201+ capillary blood collection methods against the standard reference hematology analyzer.

The study hypothesizes that the Pronto® with DCI-mini™ sensor will approximate Hb values within ±1.0 g/dL and secondly, it will correctly classify participants as anemic or not anemic with less than 31% disagreement when compared to the standard reference hematology analyzer among children 6 to 59 months of age. Additionally, the two different HemoCue® Hb 201+ capillary blood collection methodologies will both approximate Hb values within ±1.0 g/dL and secondly, it will correctly classify participants as anemic or not anemic with less than 35% disagreement when compared to the standard reference hematology analyzer among children 6 to 59 months of age.

DETAILED DESCRIPTION:
The Hb values of 132 children, between 6 and 59 months of age will be obtained, using three different Hb assessment methods during the same assessment visit for comparison with the standard reference hematology analyzer(Sysmex KN21) results.

The purpose of the research is: 1) To evaluate the accuracy of the noninvasive Masmio Pronto® device with DCI-mini sensor in measuring Hb when compared to measuring Hb using the standard reference hematology analyzer, and 2) To evaluate the accuracy of both the HemoCue® Hb 201+ gravity and wicking methodologies of capillary blood collection against the standard reference hematology analyzer.

To validate and determine the accuracy of the Pronto® with DCI-mini™ sensor, the 132 Pronto® Hb values will be compared to the Hb values obtained by the standard reference hematology analyzer to determine if the overall average difference between measurements does not exceed 1.0g/dL.

To validate and determine the accuracy of each of the two HemoCue® 201+ blood collection methods, 50% of the children will have their Hb measured using the wicking method and 50% will have their Hb measured using the gravity method. The Hb values obtained by the two different HemoCue® 201+ blood collection methods will be compared to the standard reference hematology analyzer to determine if the overall average difference between each method and the standard reference is within 1.0g/dL.

For each child, study nurse/coordinator will: collect health information from the child, categorize skin pigmentation using the Massey and Martin NIS Skin Color Scale, measure and record finger diameter using the Masimo finger measuring tool (if none of the fingers are the appropriate size for the sensor, then the big toe will be measured and used instead). Capillary blood samples of the children will be taken via finger pricking of the third or fourth digit. If a child of 6-11 months is acutely malnourished (as determined by their weight-for-height Z score), the blood drop will be obtained from their heel in accordance with Hemocue® 201+ protocol and to ensure the finger bone is not injured due to insufficient finger padding. For both blood sampling locations, the first two drops of blood will be wiped away and only the third blood drop will be used. The randomization process and the data analysis phase will not be blinded.

To determine the accuracy of the noninvasive device, the difference between Hb values obtained from the Pronto® with DCI-mini™ sensory and standard reference hematology analyzer (Sysmex KN21™) will be calculated for each child and an average obtained. In addition to the mean difference (bias), the standard deviation, 95% confidence interval, range, and limits of agreement will also be obtained. Accuracy of Hb measurement by the noninvasive device will be assessed by determining whether the measurement obtained with each noninvasive device falls within ±1.0 g/dL of the standard reference. With 100 samples and assuming the correlation between measurement methods is at least 0.93, we have 97-99% power to confirm that the average difference between the two Hb measurement methods does not exceed 1.0 g/dL. This analysis will be conducted using a paired t-test since we will be testing a limit on the difference between the measures. The prevalence rate of anemia will also be estimated for the group from the noninvasive measurements in comparison to the standard reference measurements and analyzed by paired t-test. For this comparison, our sample size of 100 affords us enough power to determine if participants are correctly classified as anemic or not anemic, with less than 31% disagreement.

A similar process will be followed for each of the two HemoCue® Hb 201+ capillary blood collection methodologies in comparison to the standard reference hematology analyzer using a paired t-test to test the limit on the difference between measures. With 50 samples and assuming the correlation between measurement methods is at least 0.93, we again have 77-99% power to confirm that the average difference between each of the two Hb measurement methods and the standard reference does not exceed 1.0 g/dL. The prevalence rate of anemia will also be estimated for each of the HemoCue® 201+ study arms for comparison with the standard reference measurements and analyzed by paired t-test. For this comparison, our sample size of 100 enables us to test if participants are correctly classified as anemic or not anemic, with less than 35% disagreement.

ELIGIBILITY:
Inclusion Criteria:

* Children, 6 to 59 months of age, receiving outpatient health care from CHUK who will already be providing a venous blood sample for their care. Outpatients typically receive care for upper respiratory infections, pneumonia, malaria, HIV infection, allergies, simple diarrhea, ear infection, malnutrition, and chronic fever. Children experiencing these health issues can be included in the sample. Children experiencing more mild health issues will also be included in the sample.
* Ability and willingness of study participant's parent/legal guardian to provide informed consent.
* Giving a venous blood sample for Hb measurement as part of their standard of care.

Exclusion Criteria:

* Younger than 6 months of age.
* Older than 59 months of age.
* Weight less than 3 kg.
* Weight greater than 30 kg.
* Any medical condition that would interfere with participant's ability to participate in the study. Such medical conditions include trauma, dehydration, shock, and all acute illnesses requiring urgent care.
* Skin abnormalities (e.g., burns, scar tissue, infections) at the planned application sites that would interfere with or preclude sensor placement and ability to transluminate the finger.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be children 6 to 59 months of age, receiving outpatient care from Centre Hospitalier Universitaire de Kigali (CHUK) and providing a venous blood sample for their health care.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pronto® Hb measurement | Day 1
  Average difference (correlation and concordance) between Hb measurements obtained using the Pronto® with DCI-mini™ sensors and the standard reference hematology analyzer, and t-test statistic.

SECONDARY OUTCOMES:
HemoCue® Hb measurement | Day 1
  Average difference (correlation and concordance) between each of the HemoCue® Hb 201+ capillary blood collection methods and the standard reference hematology analyzer, and t-test statistic.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Parker, MSc, PhD, Principal Investigator — PATH
Locations (1):
- Centre Hospitalier Universitaire de Kigali, Kigali, Rwanda